CLINICAL TRIAL: NCT04939181
Title: Efficacy of Non-invasive Neuromodulation NESA in Neuroefficiency in Basketball Players on the Field
Brief Title: Non-invasive Neuromodulation NESA in Neuroefficiency in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NESABarça
Record Dates: First submitted 2021-06-08; First posted 2021-06-25 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Basketball Player
Keywords: physical therapy modality; Electric Stimulation Therapy; basketball

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Placebo Comparator): Placebo microcurrents Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Placebo Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 10 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7. Characteristics of microcurrents:
  pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 mV and intensity 0.5 μA.
  Arms: Non-invasive Neuromodulation
Device: Placebo Non-invasive Neuromodulation — The same protocol described for the experimental group will be applied, but microcurrents device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents.
  Arms: Placebo Non-invasive Neuromodulation

SUMMARY:
Competitive team sports calendars are becoming increasingly compressed, generating changes in the effort-recovery cycle. Given this new situation, it seems necessary to analyze how it affects the physiological and performance level of semi-professional players, as well as how to observe if the non-invasive neuromodulation technique NESA helps the neuroefficiency and concentration values of said players.

DETAILED DESCRIPTION:
The design of this study is a randomised, triple blind clinical trial with placebo control.

The general configuration of the study consists of capturing the second basketball team of FC BARCELONA. For this, a double-blind capture system will be available (neither the specialist nor those responsible for recovery will know which patients are entering the complementary treatment) and two NESA XSIGNAL® devices operating in double-blind (due to the imperceptivity of the stimulation performed, there will be a placebo machine and another that applies the treatment).

At the end of the study, the results obtained between the different groups of patients will be able to be compared; those additionally treated with a device, those treated with a placebo device and those in the standard rehabilitation procedure without a device.

The variables of the study will be collected at three time points: before the intervention, during the intervention and at the end of the intervention.

The statistical analysis will be an intention-to-treat analysis. For the main outcomes variables a two factor ANOVA will-be performed (intervention-time) with a post-hoc analysis with kruskal wallis correction correction. Statistical significance will be defined as p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the team
* Participants do not present injury or pathology during the study
* In normal conditions and mentally competent to participate in the study.
* In condition to complete the study questionnaires.

Exclusion Criteria:

* Present some of the contraindications for a treatment with non-invasive neuromodulation: pacemakers, internal bleeding, do not apply electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and / or electricity phobia.
* Not having signed the informed consent.
* Present any injury or pathology during the study

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A men's basketball team will be evaluated
Enrollment: 12 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Changes in creatinine kinase level | 48 hours before the first match, immediately after the match and 48 hours after the match
  For the analysis of these biomarkers, a saliva sample, collected with Salivette containers will be necessary. Once the sample is obtained, it will be kept following the necessary security protocols and sent to a laboratory for further analysis.

SECONDARY OUTCOMES:
Kinematic demand parameters (external load) I | Through study completion, an average of 6 weeks
  Total distance traveled (meters minute)
Kinematic demand parameters (external load) II | During the match and all the intervention ( 6 weeks)
  Player Load (vector magnitude expressed as the square root of the sum of the squared instantaneous rates of change in acceleration in each of the 3 planes divided by 100) in arbitrary units (>0.02 AU; m·min-1)
Kinematic demand parameters (external load) III | During all the intervention ( 6 weeks)
  High-speed running absolute (HSR distance covered above 18 km·h -1; m·min-1
Kinematic demand parameters (external load) IV | Through study completion, an average of 6 weeks
  Relative high-speed running (RHSR, distance covered above 85% of individual maximum speed recorded in training sessions or matches; m·min-1)
Cardiovascular parameters: heart rate variability (VHR) | Up to 6 weeks
  It is proposed to observe the changes or adaptations presented by the player once the sporting activity has ceased, by quantifying the modulation between the sympathetic and parasympathetic systems
Perceptual parameters | Up to 6 weeks
  A Wellness questionnaire consisting of four questions on the level of fatigue, stress, sleep and muscle pain before the game. Each question is scored individually with scores ranging from 1 ("Very, very low or good") to 7 ("Very, very high or bad"). The higher the score, the worse the results. The largest value would be 49, while the smallest would be 4
Perceptual parameters II | During all the intervention. Up to 6 weeks
  Perception of Effort questionnaire to value perceived by the athlete will be recorded during the days of the intervention.also known as the Borg scale of perceived exertion measures the entire range of exertion that the individual perceives when exercising. The instrument consists of a table with numbers between 20 and 6, placed vertically and accompanied by qualitative evaluations between very, very strong and very, very light.

OTHER OUTCOMES:
Basketball free throw efficiency | Up to 6 weeks
  Variable analyzed by counting the number of free throws taken and the number of shots that enter the ring. To measure this type of throw during training, a protocolized Task will be carried out where each player shoots between 4 and 6 free throws (in series of 2) each training in a pressure context.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez-Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Aníbal Báez-Suárez, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Impellizzeri FM, Marcora SM, Coutts AJ. Internal and External Training Load: 15 Years On. Int J Sports Physiol Perform. 2019 Feb 1;14(2):270-273. doi: 10.1123/ijspp.2018-0935. Epub 2019 Jan 6. PMID 30614348
- [Result] Vanrenterghem J, Nedergaard NJ, Robinson MA, Drust B. Training Load Monitoring in Team Sports: A Novel Framework Separating Physiological and Biomechanical Load-Adaptation Pathways. Sports Med. 2017 Nov;47(11):2135-2142. doi: 10.1007/s40279-017-0714-2. PMID 28283992
- [Result] Kellmann M, Bertollo M, Bosquet L, Brink M, Coutts AJ, Duffield R, Erlacher D, Halson SL, Hecksteden A, Heidari J, Kallus KW, Meeusen R, Mujika I, Robazza C, Skorski S, Venter R, Beckmann J. Recovery and Performance in Sport: Consensus Statement. Int J Sports Physiol Perform. 2018 Feb 1;13(2):240-245. doi: 10.1123/ijspp.2017-0759. Epub 2018 Feb 19. PMID 29345524
- [Result] Bragazzi NL, Khoramipour K, Chaouachi A, Chamari K. Toward Sportomics: Shifting From Sport Genomics to Sport Postgenomics and Metabolomics Specialties. Promises, Challenges, and Future Perspectives. Int J Sports Physiol Perform. 2020 Sep 22;15(9):1201-1202. doi: 10.1123/ijspp.2020-0648. No abstract available. PMID 32963119
- [Result] Fernandez D, Varo F, Carmona G, Reche X. Quantification of external load of elite rink hockey players in official matches. J Sports Med Phys Fitness. 2020 Dec;60(12):1520-1525. doi: 10.23736/S0022-4707.20.11097-1. Epub 2020 Jun 30. PMID 32608935
- [Result] Torreno N, Munguia-Izquierdo D, Coutts A, de Villarreal ES, Asian-Clemente J, Suarez-Arrones L. Relationship Between External and Internal Loads of Professional Soccer Players During Full Matches in Official Games Using Global Positioning Systems and Heart-Rate Technology. Int J Sports Physiol Perform. 2016 Oct;11(7):940-946. doi: 10.1123/ijspp.2015-0252. Epub 2016 Aug 24. PMID 26816391
- [Result] Rabbani A, Clemente FM, Kargarfard M, Chamari K. Match Fatigue Time-Course Assessment Over Four Days: Usefulness of the Hooper Index and Heart Rate Variability in Professional Soccer Players. Front Physiol. 2019 Feb 19;10:109. doi: 10.3389/fphys.2019.00109. eCollection 2019. PMID 30837890
- [Result] Dong JG. The role of heart rate variability in sports physiology. Exp Ther Med. 2016 May;11(5):1531-1536. doi: 10.3892/etm.2016.3104. Epub 2016 Feb 23. PMID 27168768
- [Result] Rave G, Zouhal H, Boullosa D, Doyle-Baker PK, Saeidi A, Abderrahman AB, Fortrat JO. Heart Rate Variability is Correlated with Perceived Physical Fitness in Elite Soccer Players. J Hum Kinet. 2020 Mar 31;72:141-150. doi: 10.2478/hukin-2019-0103. eCollection 2020 Mar. PMID 32269655
- [Result] Castro-Sepulveda M, Cancino J, Fernandez-Verdejo R, Perez-Luco C, Jannas-Vela S, Ramirez-Campillo R, Del Coso J, Zbinden-Foncea H. Basal Serum Cortisol and Testosterone/Cortisol Ratio Are Related to Rate of Na+ Lost During Exercise in Elite Soccer Players. Int J Sport Nutr Exerc Metab. 2019 Nov 1;29(6):658-663. doi: 10.1123/ijsnem.2019-0129. PMID 31629352
- [Derived] Garcia F, Fernandez D, Vazquez-Guerrero J, Font R, Moreno-Planas B, Alamo-Arce D, Medina-Ramirez R, Mallol-Soler M. Recovery of the physiological status in professional basketball players using NESA neuromodulation treatment during different types of microcycles in season: A preliminary randomized clinical trial. Front Physiol. 2022 Nov 22;13:1032020. doi: 10.3389/fphys.2022.1032020. eCollection 2022. PMID 36483295